CLINICAL TRIAL: NCT06078397
Title: Remote Programming for Deep Brain Stimulation in Parkinson's Disease: a Randomized Controlled Study
Brief Title: Remote Programming for Deep Brain Stimulation in Parkinson's Disease.
Acronym: REPRO-PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RPDBSPD
Record Dates: First submitted 2023-09-20; First posted 2023-10-11 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-08

CONDITIONS: Deep Brain Stimulation; Parkinson Disease
Keywords: telemedicine; remote programming
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the Remote Programming (RP) group (Experimental): After implantation of DBS and train for RP in hospital, regularly receive RP instead of in-visit SP for parameter adjustment in 1, 3, 6 month after surgery
  Interventions: Device: remote programming
- the Standard Programming (SP) group (Active Comparator): After implantation of DBS, regularly receive SP for parameter adjustment in 1, 3, 6 month after surgery
  Interventions: Device: standard programming

INTERVENTIONS:
Device: remote programming — Remote programming (RP) is a new type of patient management method after DBS surgery, which allows physicians to understand the patient's movement symptoms and adjust parameters through video conferencing. At the same time, the RP system also includes device checks, medication adjustments, psychological counseling, and other contents. Compared to standard programming that requires going to the hospital, the application of RP can save the burden on patients and their caregivers.
  Arms: the Remote Programming (RP) group
Device: standard programming — Programming refers to a series of methods that set the parameters of the IPG after the implantation of DBS, and adjust the device parameters based on the patient's symptoms during subsequent follow-up to maintain the efficacy of electrical stimulation.
  Arms: the Standard Programming (SP) group

SUMMARY:
This study aims to conduct a randomized controlled study to compare the efficacy of remote programming (RP) on the improvement of motor function after DBS surgery in PD patients with standard programming (SP).

DETAILED DESCRIPTION:
This is a randomized controlled trial aiming at comparing the efficacy of RP and SP in post-operative management of PD patients with DBS. Enrolled patients will be randomly assigned to the RP or SP groups before surgery. After recording baseline data, regular programming sessions will be conducted through RP or SP. Patients will be followed up in 6 months after implantation, with the main goal of the differences in motor symptom improvement between the two groups and the secondary goal of the difference in safety and economic benefits between both methods.

ELIGIBILITY:
Inclusion Criteria:

1. Adult primary Parkinson's disease patients who meet the diagnostic criteria for Parkinson's disease in China (2016 edition), aged 18-75 years
2. Comply with the surgical indications of the "Expert Consensus on Deep Brain Stimulation Therapy for Parkinson's Disease in China (Second Edition)" and complete bilateral STN-DBS surgery
3. Accurate lead position verified by postoperative CT examination
4. The implanted DBS device has remote programming function
5. Having an internet connection at home or in the area that will receive remote postoperative management, and being able to participate in remote symptom assessment and remote programming
6. Able to communicate fluently, and after education, I and my caregivers are proficient in using the patient client of the remote program control system
7. Understand potential risks/benefits, agree to participate in the study, study procedures, agree to complete the study follow-up, and comply with the requirements of the study protocol.

Exclusion Criteria:

1. The preoperative concise mental state examination (MMSE) score of DBS indicates moderate or above cognitive impairment
2. Severe complications after DBS surgery, such as stroke, encephalitis, wound infection, etc.
3. Lack of cooperation, or inability to understand the experimental plan or provide informed consent for any reason
4. Unable to provide stable network signal or unable to provide 4 × 1.5 m space for motion evaluation
5. Other researchers believe that factors may not be suitable for research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The unified Parkinson's disease rating scale (UPDRS) Part III | Preoperation and 6 months after surgery
  The unified Parkinson's disease rating scale (UPDRS) Part III is made up of motor examinations (18 items). Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). Score range: 0-132, 32 and below is mild, 59 and above is severe.
Cost-effectiveness | 6 months after surgery
  Quality Adjusted Life Years estimated by the cost and EQ-5D-3L.

SECONDARY OUTCOMES:
The unified Parkinson's disease rating scale (UPDRS) Part I, II and IV. | Preoperation and 6 months after surgery.
  The unified Parkinson's disease rating scale (UPDRS) is made up of these sections:
  Part I: Nonmotor experiences of daily living: 13 items. Score range: 0-52, 10 and below is mild, 22 and above is severe.
  Part II: Motor experiences of daily living: 13 items. Score range: 0-52, 12 and below is mild, 30 and above is severe.
  Part III: Motor examinations :18 items. Score range: 0-132, 32 and below is mild, 59 and above is severe.
  Part IV: Motor complications: 6 items. Score range: 0-24, 4 and below is mild, 13 and above is severe.
  Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe).
Parkinson's Disease Questionaire-8 (PDQ-8) | Preoperation and 6 months after surgery.
  The Parkinson's Disease Questionaire-8 (PDQ-8) is an eight-question instrument with questions taken from each domain of 39-item Parkinson's Disease Questionnaire (PDQ-39). Each question is scored between 0 and 4, higher scores indicate poorer quality of life.
European Quality of Life 5 Dimensions 3 Level Version | Preoperation and 6 months after surgery.
  The European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Beck Depression Inventory (BDI-II) | Preoperation and 6 months after surgery.
  The Beck Depression Inventory (BDI-II) is a widely used 21-item self-report inventory measuring the severity of depression in adolescents and adults. Each item is scored between 0 and 3, a score of 10 to 18 indicates mild depression, and 30 or above indicates severe depression.
Beck Anxiety Inventory (BAI) | Preoperation and 6 months after surgery.
  Beck Anxiety Inventory (BAI) is a self-report inventory measuring 21 common somatic and cognitive symptoms of anxiety. Each item is scored by a Likert scale ranging from 0 to 3 and raw scores ranging from 0 to 63, classified as minimal anxiety (0 to 7), mild anxiety (8 to 15), moderate anxiety (16 to 25), and severe anxiety (30 to 63).
Mini-Mental State Examination (MMSE) | Preoperation and 6 months after surgery.
  A Mini-Mental State Examination (MMSE) is a set of 11 questions with scores ranging from 0~30 points used to check for cognitive impairment (problems with thinking, communication, understanding and memory). Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Cost of patients' perspective | 6 months after surgery.
  Costs of patients and caregivers' perspective were taken into account: a.travel, b. informal care and c. income loss (calculated by time). Costs was collected by unified questionnaires.
Telehealth Satisfaction Survey (TeSS) | Collected within 2 days (48 hours) after each programming.
  Telehealth Satisfaction Survey (TeSS) is a 10-item scale for Satisfaction scores on the, Each response was rated as poor, fair, good and excellent (0 to 3). Higher scores indicated higher satisfaction with telehealth.
The Patient Global Impression of Change (PGIC) | Collected within 2 days (48 hours) after each programming.
  The Patient Global Impression of Change (PGIC) scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Safety: Rate of programming related adverse events | Collected within 2 days (48 hours) after each programming.
  The adverse events questionnaire is composed of 3 parts: 1.Hardware related (eg. Poor Internet connection); 2. Operation related (eg. Low battery of devices); 3.Stimulation related (eg. Dyskinesia after programming); 4. Others.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No